CLINICAL TRIAL: NCT06019234
Title: Uvenile Systemic Sclerosis, a Retrospective Epidemiological Study on a French Cohort
Brief Title: Juvenile Systemic Sclerosis, a Retrospective Epidemiological Study on a French Cohort
Acronym: JSSc
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9028
Record Dates: First submitted 2023-08-24; First posted 2023-08-31 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-08

CONDITIONS: Juvenile Systemic Sclerosis
Keywords: Systemic Sclerosis; Juvenile Systemic Sclerosis; Immunosuppressive treatments
MeSH Terms: conditions — Juvenile systemic scleroderma; Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Scleroderma is an inflammatory attack of the vessels leading to localized or multisystemic sclerosis. It is a rare autoimmune pathology in pediatrics.

The incidence in pediatrics is very low (about 4 per million according to an American) and therefore the data on the pathology very poor, especially on the therapeutic level.

The proposed immunosuppressive treatments are extrapolated from data in adults. The evolution of connectivity does not seem quite identical to the evolution of adult scleroderma, adaptation of treatments seems judicious. However, data on the evolution under therapy in children are still poor.

Complications related to the pathology, iatrogeny and diagnostic delay are the first causes of mortality from this pathology and deserve to be studied and if possible avoided.

The main hypothesis of the research being to bring together the experiences of the various reference and competence centers in France concerning the clinical presentation, management and follow-up of children with systemic sclerosis.

ELIGIBILITY:
Inclusion criteria:

* Minor subject (<18 years old)
* Diagnosis of systemic sclerosis between 01/01/2012 and 30/06/2022.
* Subject (and/or his parental authority) who has not expressed, after being informed, his opposition to the reuse of his data for the purposes of this research.

Exclusion criteria:

- Subject (or his parents) having expressed his (their) opposition to participating in the study

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Minor subject (<18 years old) having a systemic sclerosis between 01/01/2012 and 30/06/2022.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2024-10-03 (Estimated); Study Completion 2024-10-03 (Estimated)

PRIMARY OUTCOMES:
The therapeutic response was evaluated by the EULAR DAS 28 -CRP | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ariane ZALOSZYC, MD, Study Director — University Hospitals of Strasbourg
Locations (1):
- Service de Pédiatrie 1 - CHU de Strasbourg - France, Strasbourg, France